CLINICAL TRIAL: NCT04826003
Title: An Open-Label, Multicenter, Phase Ib Study To Evaluate Safety, Pharmacokinetics, Pharmacodynamics, And Preliminary Anti-Tumor Activity Of RO7122290, A Fibroblast Activation Protein-A (FAP) Targeted 4-1BB Ligand (CD137L), In Combination With Cibisatamab With Obinutuzumab Pre-Treatment, In Participants With Previously Treated, Metastatic, Microsatellite-stable Colorectal Adenocarcinoma With High CEACAM5 Expression
Brief Title: Study To Evaluate Safety, Pharmacokinetics, Pharmacodynamics, And Preliminary Anti-Tumor Activity Of RO7122290 In Combination With Cibisatamab With Obinutuzumab Pre-Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP42675
Record Dates: First submitted 2021-03-16; First posted 2021-04-01 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Microsatellite stable;; Metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — cibisatamab; obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part I: Dose-escalation of RO7122290 (Experimental): The dose-escalation of RO7122290 will use a QW dosing schedule of RO7122290 in combination with a Q3W dosing interval for cibisatamab with obinutuzumab pre-treatment. The starting dose for RO7122290 will be 35 mg, which represents the human equivalent dose for the minimal pharmacologically active dose (1 mg/kg) in mice.
  Interventions: Drug: RO7122290; Drug: Cibisatamab; Drug: Obinutuzumab
- Part II: Dose-expansion of RO7122290 (Experimental): Part II of this study will evaluate selected dose levels of RO7122290 from Part I (a QW RO712290 administration in combination with a Q3W cibisatamab administration with obinutuzumab pre-treatment) in a Q3W regimen in combination with a Q3W cibisatamab administration with obinutuzumab pre-treatment.
  Interventions: Drug: RO7122290; Drug: Cibisatamab; Drug: Obinutuzumab

INTERVENTIONS:
Drug: RO7122290 — RO7122290 will be administered using a QW (Part I) or Q3W (Part I or Part II) schedule in combination with 100 mg cibisatamab Q3W with obinutuzumab pre-treatment. The maximum dose of RO7122290 to be explored in combination with cibisatamab with obinutuzumab pre-treatment in this study is 500 mg for the QW dosing interval (Part I) or 1500 mg for the Q3W dosing interval (Part I or Part II).
Drug: Cibisatamab — Cibisatamab will be administered to participants at a fixed dose of 100 mg Q3W (100 mg on Day 1 of each 21-day cycle).
Drug: Obinutuzumab — Obinutuzumab will be administered (IV) as pre-treatment on Day - 8/- 7 (split dose) or
  - 8 (single dose) prior to C1D1 of cibisatamab and as re-treatment every 6 months if the participant is still receiving cibisatamab

SUMMARY:
This is an open-label, multicenter, Phase Ib study to determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) in the weekly (QW) and/or every 3 weeks (Q3W) regimens, safety, tolerability, PK, immunogenicity, PD profile and to evaluate preliminary anti-tumor activity of RO7122290 in combination with cibisatamab Q3W after pretreatment with obinutuzumab, in participants with previously treated metastatic, microsatellite-stable colorectal adenocarcinoma with high CEACAM5 expression

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma originating from the colon or rectum.
* Metastatic disease (Stage IV American Joint Committee on Cancer, Version 7) not amenable to local treatment.
* Tumors that are MSS (microsatellite-stable) or MSI-low (microsatellite instable low), as determined by a certified laboratory
* Participants with tumors that have high CEACAM5 expression as determined by qRT-PCR in an archival tumor sample or if not available, in a fresh tumor biopsy and documented through central testing of a representative tumor tissue specimen performed at baseline
* Experienced disease progression during or within 3 months following the last administration of approved standard therapies.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Life expectancy of ≥12 weeks
* Adequate organ functions.
* Serum creatinine within normal limits or a calculated glomerular filtration rate of ≥ 60 mL/min/1.73 m2 for participants with serum creatinine levels above or below the institutional normal value.
* Serum albumin ≥30 g/L (3.0 g/dL).
* Lactate dehydrogenase ≤ 2.5 x ULN.
* Adequate contraception

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.
* History of leptomeningeal disease
* Non-irradiated tumor lesions > 2 cm at critical sites (e.g., paraspinal, paratracheal, mediastinal, precarnial, sub-glottal) where tumor swelling induced by cibisatamab is expected to lead to significant complications. Irradiation must be completed at least 14 days prior to initiation of study treatment.
* Dyspnea or peripheral capillary oxygen saturation < 92% at rest at baseline for patients with bilateral lung lesions or metastases in the remaining lung following lobectomy or pneumonectomy
* Pleural effusion requiring drainage procedures.
* Pleural effusion and/or pleural lesions involving both lungs
* Active interstitial lung disease (ILD), pneumonitis, or a history of ILD/pneumonitis requiring treatment with steroids or history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Severe dyspnea at rest due to complications of advanced malignancy or requiring supplementary oxygen therapy.
* Patients with > 10 bilateral pulmonary lesions
* Patients with pulmonary miliary metastatic pattern (innumerable small lesions) or pulmonary lymphangitic carcinomatosis.
* Significant cardiovascular/cerebrovascular disease within 6 months prior to Day 1 of study drug administration
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 2 weeks prior to initiation of study treatment.
* History of progressive multifocal leukoencephalopathy
* Uncontrolled tumor-related pain.
* Uncontrolled ascites requiring recurrent drainage procedures (QW or more frequently). Participants with indwelling catheters are allowed.
* Patients with pericardial effusion.
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis for a more comprehensive list of autoimmune diseases and immune deficiencies).
* Active tuberculosis that has required treatment within 3 years prior to initiation of study treatment or latent tuberculosis that has not been appropriately treated.
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study.
* History of malignancy other than CRC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including diabetes mellitus, history of relevant pulmonary disorders, or other disease with ongoing fibrosis (such as scleroderma, pulmonary fibrosis, emphysema, neurofibromatosis, palmar/plantar fibromatosis).
* Known active infection, or reactivation of a latent infection, whether bacterial, viral (including, but not limited to, Epstein-Barr virus infection), fungal, mycobacterial, or other pathogens (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization or treatment with systemic antibiotics (IV and oral antibiotic treatment must have been completed at least 4 and 2 weeks, respectively, prior to initiation of study treatment).
* Prior allogeneic stem cell or solid organ transplantation.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment.
* History of chronic liver disease or evidence of hepatic cirrhosis.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that give reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug.
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy and to chimeric or humanized antibodies or fusion proteins.
* Major surgery or significant traumatic injury < 28 days prior to the first obinutuzumab infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment.
* Treatment with any systemic anti-cancer therapy, including chemotherapy or hormonal therapy, within 28 days prior to initiation of study treatment
* Prior treatment with T-cell bispecifics (TCBs), CD137 (4-1BB) agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies, unless discussed and agreed by the Sponsor.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2) within 4 weeks or 5 half-lives (whatever if longer) prior to initiation of study treatment.
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment.
* Adverse events from prior anti-cancer therapy that have not resolved to Grade 1 or better with the exception of alopecia of any grade and Grade ≤ 2 peripheral neuropathy.
* Known hypersensitivity to Chinese hamster ovary cell products.
* Known allergy or hypersensitivity to any of the study drugs or any of their excipients.
* Any participant actively taking anti platelet medication (aspirin, clopidogrel, ticagrelor, etc.) or any participant who is fully anti coagulated with warfarin, low molecular weight heparin or a novel oral anti-coagulant including dabigatran, rivaroxaban, epixaban, etc.
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Part I: Occurrence of dose-limiting toxicities | Baseline up to 21 days
  The DLT observation period is defined as a period of 21 days after the first administration of RO7122290 combined with cibisatamab. Additional days (maximum 3 days per dosing) are allowed in case of treatment delays for non-safety reasons.
  Participants are evaluable for DLT assessment, if they have received one dose of cibisatamab and at least two doses of RO7122290 during the DLT period.
Percentage of Participants with Adverse Events | Baseline up to 28 months
  Incidence, nature, and severity of adverse events (AEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5 with the exception of cytokine release syndrome (CRS), which is graded according to the ASTCT grading scale for CRS (with individual signs and symptoms of CRS graded separately using the CTCAE v5.0 grading scale)

SECONDARY OUTCOMES:
Serum concentration of RO7122290 over time | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1: Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); Day 4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose), D9 (24h postdose); D12 (96h postdose); D15 (Predose, 15 minutes, 4h postdose); D16 (24h postdose); Cycle 2 Day 1 (Predose, 15 minutes postdose); D2 (24h postdose), D8 (Predose, 15 minutes, 4h postdose); D9 (24h postdose); D15 (Predose, 15 minutes postdose); Subsequent Cycles D1 (Predose, 15 minutes postdose); D8 (Predose, 15 minutes postdose); D15 ((Predose, 15 minutes postdose); Discontinuation visit; 28 Day Safety Follow Up Visit, 90 (±7 days) post last dose after last dose of RO7122290.
  Part II:
  Cycle 1 Day 1 (Predose, 15minutes 4h, 8h, postdose); Day 2; D4; D8; D9; D12 ; D15; Cycle 2, Day 1 (Predose, 15 minutes postdose); Day 2; D8; D9; D12; Subsequent Cycles Day 1 (Predose, 15 minutes postdose) D8; D16; Discontinuation visit; 28 Day Follow Up; Safety FU Visit. Each cycle is 21 days
Plasma concentration of RO7122290 over time | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1: Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); Day 4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose), D9 (24h postdose); D12 (96h postdose); D15 (Predose, 15 minutes, 4h postdose); D16 (24h postdose); Cycle 2 Day 1 (Predose, 15 minutes postdose); D2 (24h postdose), D8 (Predose, 15 minutes, 4h postdose); D9 (24h postdose); D15 (Predose, 15 minutes postdose); Subsequent Cycles D1 (Predose, 15 minutes postdose); D8 (Predose, 15 minutes postdose); D15 ((Predose, 15 minutes postdose); Discontinuation visit; 28 Day Safety Follow Up Visit, 90 (±7 days) post last dose after last dose of RO7122290.
  Part II:
  Cycle 1 Day 1 (Predose, 15minutes 4h, 8h, postdose); Day 2; D4; D8; D9; D12 ; D15; Cycle 2, Day 1 (Predose, 15 minutes postdose); Day 2; D8; D9; D12; Subsequent Cycles Day 1 (Predose, 15 minutes postdose) D8; D16; Discontinuation visit; 28 Day Follow Up; Safety FU Visit. Each cycle is 21 days
Maximum concentration (Cmax) of RO7122290 | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1: Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); Day 4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose), D9 (24h postdose); D12 (96h postdose); D15 (Predose, 15 minutes, 4h postdose); D16 (24h postdose); Cycle 2 Day 1 (Predose, 15 minutes postdose); D2 (24h postdose), D8 (Predose, 15 minutes, 4h postdose); D9 (24h postdose); D15 (Predose, 15 minutes postdose); Subsequent Cycles D1 (Predose, 15 minutes postdose); D8 (Predose, 15 minutes postdose); D15 ((Predose, 15 minutes postdose); Discontinuation visit; 28 Day Safety Follow Up Visit, 90 (±7 days) post last dose after last dose of RO7122290.
  Part II:
  Cycle 1 Day 1 (Predose, 15minutes 4h, 8h, postdose); Day 2; D4; D8; D9; D12 ; D15; Cycle 2, Day 1 (Predose, 15 minutes postdose); Day 2; D8; D9; D12; Subsequent Cycles Day 1 (Predose, 15 minutes postdose) D8; D16; Discontinuation visit; 28 Day Follow Up; Safety FU Visit. Each cycle is 21 days
Time of maximum concentration (Tmax) of RO7122290 | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1: Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); Day 4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose), D9 (24h postdose); D12 (96h postdose); D15 (Predose, 15 minutes, 4h postdose); D16 (24h postdose); Cycle 2 Day 1 (Predose, 15 minutes postdose); D2 (24h postdose), D8 (Predose, 15 minutes, 4h postdose); D9 (24h postdose); D15 (Predose, 15 minutes postdose); Subsequent Cycles D1 (Predose, 15 minutes postdose); D8 (Predose, 15 minutes postdose); D15 ((Predose, 15 minutes postdose); Discontinuation visit; 28 Day Safety Follow Up Visit, 90 (±7 days) post last dose after last dose of RO7122290.
  Part II:
  Cycle 1 Day 1 (Predose, 15minutes 4h, 8h, postdose); Day 2; D4; D8; D9; D12 ; D15; Cycle 2, Day 1 (Predose, 15 minutes postdose); Day 2; D8; D9; D12; Subsequent Cycles Day 1 (Predose, 15 minutes postdose) D8; D16; Discontinuation visit; 28 Day Follow Up; Safety FU Visit. Each cycle is 21 days
Clearance (CL) of RO7122290 | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1: Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); Day 4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose), D9 (24h postdose); D12 (96h postdose); D15 (Predose, 15 minutes, 4h postdose); D16 (24h postdose); Cycle 2 Day 1 (Predose, 15 minutes postdose); D2 (24h postdose), D8 (Predose, 15 minutes, 4h postdose); D9 (24h postdose); D15 (Predose, 15 minutes postdose); Subsequent Cycles D1 (Predose, 15 minutes postdose); D8 (Predose, 15 minutes postdose); D15 ((Predose, 15 minutes postdose); Discontinuation visit; 28 Day Safety Follow Up Visit, 90 (±7 days) post last dose after last dose of RO7122290.
  Part II:
  Cycle 1 Day 1 (Predose, 15minutes 4h, 8h, postdose); Day 2; D4; D8; D9; D12 ; D15; Cycle 2, Day 1 (Predose, 15 minutes postdose); Day 2; D8; D9; D12; Subsequent Cycles Day 1 (Predose, 15 minutes postdose) D8; D16; Discontinuation visit; 28 Day Follow Up; Safety FU Visit. Each cycle is 21 days
Volume of distribution (V) of RO7122290 | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1: Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); Day 4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose), D9 (24h postdose); D12 (96h postdose); D15 (Predose, 15 minutes, 4h postdose); D16 (24h postdose); Cycle 2 Day 1 (Predose, 15 minutes postdose); D2 (24h postdose), D8 (Predose, 15 minutes, 4h postdose); D9 (24h postdose); D15 (Predose, 15 minutes postdose); Subsequent Cycles D1 (Predose, 15 minutes postdose); D8 (Predose, 15 minutes postdose); D15 ((Predose, 15 minutes postdose); Discontinuation visit; 28 Day Safety Follow Up Visit, 90 (±7 days) post last dose after last dose of RO7122290.
  Part II:
  Cycle 1 Day 1 (Predose, 15minutes 4h, 8h, postdose); Day 2; D4; D8; D9; D12 ; D15; Cycle 2, Day 1 (Predose, 15 minutes postdose); Day 2; D8; D9; D12; Subsequent Cycles Day 1 (Predose, 15 minutes postdose) D8; D16; Discontinuation visit; 28 Day Follow Up; Safety FU Visit. Each cycle is 21 days
Area under the curve (AUC) of RO7122290 | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1: Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); Day 4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose), D9 (24h postdose); D12 (96h postdose); D15 (Predose, 15 minutes, 4h postdose); D16 (24h postdose); Cycle 2 Day 1 (Predose, 15 minutes postdose); D2 (24h postdose), D8 (Predose, 15 minutes, 4h postdose); D9 (24h postdose); D15 (Predose, 15 minutes postdose); Subsequent Cycles D1 (Predose, 15 minutes postdose); D8 (Predose, 15 minutes postdose); D15 ((Predose, 15 minutes postdose); Discontinuation visit; 28 Day Safety Follow Up Visit, 90 (±7 days) post last dose after last dose of RO7122290.
  Part II:
  Cycle 1 Day 1 (Predose, 15minutes 4h, 8h, postdose); Day 2; D4; D8; D9; D12 ; D15; Cycle 2, Day 1 (Predose, 15 minutes postdose); Day 2; D8; D9; D12; Subsequent Cycles Day 1 (Predose, 15 minutes postdose) D8; D16; Discontinuation visit; 28 Day Follow Up; Safety FU Visit. Each cycle is 21 days
Half-life (t1/2) of RO7122290 | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1: Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); Day 4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose), D9 (24h postdose); D12 (96h postdose); D15 (Predose, 15 minutes, 4h postdose); D16 (24h postdose); Cycle 2 Day 1 (Predose, 15 minutes postdose); D2 (24h postdose), D8 (Predose, 15 minutes, 4h postdose); D9 (24h postdose); D15 (Predose, 15 minutes postdose); Subsequent Cycles D1 (Predose, 15 minutes postdose); D8 (Predose, 15 minutes postdose); D15 ((Predose, 15 minutes postdose); Discontinuation visit; 28 Day Safety Follow Up Visit, 90 (±7 days) post last dose after last dose of RO7122290.
  Part II:
  Cycle 1 Day 1 (Predose, 15minutes 4h, 8h, postdose); Day 2; D4; D8; D9; D12 ; D15; Cycle 2, Day 1 (Predose, 15 minutes postdose); Day 2; D8; D9; D12; Subsequent Cycles Day 1 (Predose, 15 minutes postdose) D8; D16; Discontinuation visit; 28 Day Follow Up; Safety FU Visit. Each cycle is 21 days
Serum concentration of Cibisatamab over time | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); D4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose); D15 (Predose); Cycle 2 Day 1 (Predose), Discontinuation visit
  Part II:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h postdose); Day 2 (24h postdose); D8 (Predose, 15 minutes, 4h postdose); Cycle 2 Day 1 (Predose, 15 min, 4h postdose,); Day 2 (24h postdose); D8 (168h postdose); C3-16 D1, then every 4th cycle (Predose); Discontinuation visit. Each cycle is 21 days
Plasma concentration of Cibisatamab over time | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); D4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose); D15 (Predose); Cycle 2 Day 1 (Predose), Discontinuation visit
  Part II:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h postdose); Day 2 (24h postdose); D8 (Predose, 15 minutes, 4h postdose); Cycle 2 Day 1 (Predose, 15 min, 4h postdose,); Day 2 (24h postdose); D8 (168h postdose); C3-16 D1, then every 4th cycle (Predose); Discontinuation visit. Each cycle is 21 days
Maximum concentration (Cmax) of Cibisatamab | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); D4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose); D15 (Predose); Cycle 2 Day 1 (Predose), Discontinuation visit
  Part II:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h postdose); Day 2 (24h postdose); D8 (Predose, 15 minutes, 4h postdose); Cycle 2 Day 1 (Predose, 15 min, 4h postdose,); Day 2 (24h postdose); D8 (168h postdose); C3-16 D1, then every 4th cycle (Predose); Discontinuation visit. Each cycle is 21 days
Time of maximum concentration (Tmax) of Cibisatamab | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); D4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose); D15 (Predose); Cycle 2 Day 1 (Predose), Discontinuation visit
  Part II:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h postdose); Day 2 (24h postdose); D8 (Predose, 15 minutes, 4h postdose); Cycle 2 Day 1 (Predose, 15 min, 4h postdose,); Day 2 (24h postdose); D8 (168h postdose); C3-16 D1, then every 4th cycle (Predose); Discontinuation visit. Each cycle is 21 days
Clearance (CL) of Cibisatamab | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); D4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose); D15 (Predose); Cycle 2 Day 1 (Predose), Discontinuation visit
  Part II:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h postdose); Day 2 (24h postdose); D8 (Predose, 15 minutes, 4h postdose); Cycle 2 Day 1 (Predose, 15 min, 4h postdose,); Day 2 (24h postdose); D8 (168h postdose); C3-16 D1, then every 4th cycle (Predose); Discontinuation visit. Each cycle is 21 days
Volume of distribution (V) of Cibisatamab | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); D4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose); D15 (Predose); Cycle 2 Day 1 (Predose), Discontinuation visit
  Part II:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h postdose); Day 2 (24h postdose); D8 (Predose, 15 minutes, 4h postdose); Cycle 2 Day 1 (Predose, 15 min, 4h postdose,); Day 2 (24h postdose); D8 (168h postdose); C3-16 D1, then every 4th cycle (Predose); Discontinuation visit. Each cycle is 21 days
Area under the curve (AUC) of Cibisatamab | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); D4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose); D15 (Predose); Cycle 2 Day 1 (Predose), Discontinuation visit
  Part II:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h postdose); Day 2 (24h postdose); D8 (Predose, 15 minutes, 4h postdose); Cycle 2 Day 1 (Predose, 15 min, 4h postdose,); Day 2 (24h postdose); D8 (168h postdose); C3-16 D1, then every 4th cycle (Predose); Discontinuation visit. Each cycle is 21 days
Half-life (t1/2) of Cibisatamab | Baseline up to 28 months (detailed time frame provided in description)
  Part I:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h, 8h postdose); Day 2 (24h postdose); D4 (72h postdose); D8 (Predose, 15 minutes, 4h postdose); D15 (Predose); Cycle 2 Day 1 (Predose), Discontinuation visit
  Part II:
  Cycle 1 Day 1 (Predose, 15 minutes, 4h postdose); Day 2 (24h postdose); D8 (Predose, 15 minutes, 4h postdose); Cycle 2 Day 1 (Predose, 15 min, 4h postdose,); Day 2 (24h postdose); D8 (168h postdose); C3-16 D1, then every 4th cycle (Predose); Discontinuation visit. Each cycle is 21 days
Serum concentration of Obinutuzumab over time | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: D -13 (Predose, 15 minutes postdose); D -12 (only in case of split dosing, done on D-13 and D-12: (Predose, 15 minutes postdose); D8 (Predose); Subsequent Cycles (Predose); Discontinuation visit. Each cycle is 21 days
Plasma concentration of Obinutuzumab over time | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: D -13 (Predose, 15 minutes postdose); D -12 (only in case of split dosing, done on D-13 and D-12: (Predose, 15 minutes postdose); D8 (Predose); Subsequent Cycles (Predose); Discontinuation visit. Each cycle is 21 days
Maximum concentration (Cmax) of Obinutuzumab | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: D -13 (Predose, 15 minutes postdose); D -12 (only in case of split dosing, done on D-13 and D-12: (Predose, 15 minutes postdose); D8 (Predose); Subsequent Cycles (Predose); Discontinuation visit. Each cycle is 21 days
Time of maximum concentration (Tmax) of Obinutuzumab | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: D -13 (Predose, 15 minutes postdose); D -12 (only in case of split dosing, done on D-13 and D-12: (Predose, 15 minutes postdose); D8 (Predose); Subsequent Cycles (Predose); Discontinuation visit. Each cycle is 21 days
Clearance (CL) of Obinutuzumab | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: D -13 (Predose, 15 minutes postdose); D -12 (only in case of split dosing, done on D-13 and D-12: (Predose, 15 minutes postdose); D8 (Predose); Subsequent Cycles (Predose); Discontinuation visit. Each cycle is 21 days
Volume of distribution (V) of Obinutuzumab | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: D -13 (Predose, 15 minutes postdose); D -12 (only in case of split dosing, done on D-13 and D-12: (Predose, 15 minutes postdose); D8 (Predose); Subsequent Cycles (Predose); Discontinuation visit. Each cycle is 21 days
Area under the curve (AUC) of Obinutuzumab | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: D -13 (Predose, 15 minutes postdose); D -12 (only in case of split dosing, done on D-13 and D-12: (Predose, 15 minutes postdose); D8 (Predose); Subsequent Cycles (Predose); Discontinuation visit. Each cycle is 21 days
Half-life (t1/2) of Obinutuzumab | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: D -13 (Predose, 15 minutes postdose); D -12 (only in case of split dosing, done on D-13 and D-12: (Predose, 15 minutes postdose); D8 (Predose); Subsequent Cycles (Predose); Discontinuation visit. Each cycle is 21 days
Percentage of Participants with RO7122290 anti-drug antibodies (ADAs) during the study relative to the prevalence of ADA at baseline | Baseline up to 28 months (detailed time frame provided in description)
  Cycle 1: Day 1, 8, 15; Cycles 3, 4, 6, 8: Day 1; Discontinuation visit. Each cycle is 21 days
Percentage of Participants with Cibisatamab anti-drug antibodies (ADAs) during the study relative to the prevalence of ADA at baseline | Baseline up to 28 months (detailed time frame provided in description)
  Cycle 1 Day 1 (Predose, 15 minutes postdose); Cycle 2 Day 1 (Predose, 15 minutes postdose); Day 8 (Predose); C3-16 D1, then every 4th cycle; Discontinuation visit. Each cycle is 21 days
Percentage of Participants with Obinutuzumab anti-drug antibodies (ADAs) during the study relative to the prevalence of ADA at baseline | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: Day -13, Day -12 (only in case of split dosing, done on D-13 and D-12); C3, 4, 6, 8 Day 1; Discontinuation visit. Each cycle is 21 days
Treatment-induced change on T-cell proliferation (CD8/Ki67) | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: day -13, Day -12 (only in case of split dosing, done on D-13 and D-12); Cycle 1, Day 1;4, 8, 9, 12, 15, 16; Cycle 2, Day 1, 2, 8, 9, 12, 15; C3-12 D1, then every 4th cycle; Discontinuation visit; 28 Day Safety Follow Up; 90 (±7 days) post last dose after last dose of RO7122290 or cibisatamab 180 (+30) days after last dose. Each cycle is 21 days
Treatment-induced change on T-cell activation (CD8/4-1BB) | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: day -13, Day -12 (only in case of split dosing, done on D-13 and D-12); Cycle 1, Day 1;4, 8, 9, 12, 15, 16; Cycle 2, Day 1, 2, 8, 9, 12, 15; C3-12 D1, then every 4th cycle; Discontinuation visit; 28 Day Safety Follow Up; 90 (±7 days) post last dose after last dose of RO7122290 or cibisatamab 180 (+30) days after last dose. Each cycle is 21 days
Treatment-induced change on tumor necrosis factor alpha (TNF-alpha) levels | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: day -13, Day -12 (only in case of split dosing, done on D-13 and D-12); Cycle 1, Day 1;4, 8, 9, 12, 15, 16; Cycle 2, Day 1, 2, 8, 9, 12, 15; C3-12 D1, then every 4th cycle; Discontinuation visit; 28 Day Safety Follow Up; 90 (±7 days) post last dose after last dose of RO7122290 or cibisatamab 180 (+30) days after last dose. Each cycle is 21 days
Treatment-induced change on interferon gamma (IFN-gamma) levels | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: day -13, Day -12 (only in case of split dosing, done on D-13 and D-12); Cycle 1, Day 1;4, 8, 9, 12, 15, 16; Cycle 2, Day 1, 2, 8, 9, 12, 15; C3-12 D1, then every 4th cycle; Discontinuation visit; 28 Day Safety Follow Up; 90 (±7 days) post last dose after last dose of RO7122290 or cibisatamab 180 (+30) days after last dose. Each cycle is 21 days
Treatment-induced change on Interleukin (IL)-2 levels | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: day -13, Day -12 (only in case of split dosing, done on D-13 and D-12); Cycle 1, Day 1;4, 8, 9, 12, 15, 16; Cycle 2, Day 1, 2, 8, 9, 12, 15; C3-12 D1, then every 4th cycle; Discontinuation visit; 28 Day Safety Follow Up; 90 (±7 days) post last dose after last dose of RO7122290 or cibisatamab 180 (+30) days after last dose. Each cycle is 21 days
Treatment-induced change on Interleukin (IL)-6 levels | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: day -13, Day -12 (only in case of split dosing, done on D-13 and D-12); Cycle 1, Day 1;4, 8, 9, 12, 15, 16; Cycle 2, Day 1, 2, 8, 9, 12, 15; C3-12 D1, then every 4th cycle; Discontinuation visit; 28 Day Safety Follow Up; 90 (±7 days) post last dose after last dose of RO7122290 or cibisatamab 180 (+30) days after last dose. Each cycle is 21 days
Treatment-induced change on Interleukin (IL)-8 levels | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: day -13, Day -12 (only in case of split dosing, done on D-13 and D-12); Cycle 1, Day 1;4, 8, 9, 12, 15, 16; Cycle 2, Day 1, 2, 8, 9, 12, 15; C3-12 D1, then every 4th cycle; Discontinuation visit; 28 Day Safety Follow Up; 90 (±7 days) post last dose after last dose of RO7122290 or cibisatamab 180 (+30) days after last dose. Each cycle is 21 days
Treatment-induced change on Interleukin (IL)-10 levels | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: day -13, Day -12 (only in case of split dosing, done on D-13 and D-12); Cycle 1, Day 1;4, 8, 9, 12, 15, 16; Cycle 2, Day 1, 2, 8, 9, 12, 15; C3-12 D1, then every 4th cycle; Discontinuation visit; 28 Day Safety Follow Up; 90 (±7 days) post last dose after last dose of RO7122290 or cibisatamab 180 (+30) days after last dose. Each cycle is 21 days
Treatment-induced change on Granulocyte-macrophage colony-stimulating factor (GM-CSF) levels | Baseline up to 28 months (detailed time frame provided in description)
  Obinutuzumab pretreatment: day -13, Day -12 (only in case of split dosing, done on D-13 and D-12); Cycle 1, Day 1;4, 8, 9, 12, 15, 16; Cycle 2, Day 1, 2, 8, 9, 12, 15; C3-12 D1, then every 4th cycle; Discontinuation visit; 28 Day Safety Follow Up; 90 (±7 days) post last dose after last dose of RO7122290 or cibisatamab 180 (+30) days after last dose. Each cycle is 21 days
Objective response rate (ORR) defined as complete response (CR) + partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline up to 28 months
  Objective response rate (ORR) is determined as the rate of participants with an objective tumor response of CR or PR. ORR will be derived for RECIST Version 1.1 and will be based on Investigators' assessment.
Disease control rate (DCR); defined as response rate (RR) + stable disease (SD) according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline up to 28 months
  Disease control rate (DCR) is determined as the rate of participants with an objective tumor response of CR, PR or SD. DCR will be derived for RECIST Version 1.1 and will be based on Investigators' assessment.
Duration of response (DoR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline up to 28 months
  DoR will be calculated for participants who have a best overall response of CR or PR and will be defined as the time from first occurrence of a documented OR until the time of documented disease progression or death (death within 30 days from last study treatment) from any cause, whichever occurs first. Censoring
Progression-free survival (PFS) according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline up to 28 months
  PFS will be defined as the time from first dose of cibisatamab or RO7122290 (C1D1) to the first occurrence of documented disease progression (based on RECIST Version 1.1 Investigator's assessment) or death from any cause, whichever occurs first. For participants who do not have documented progressive disease or death (within 30 days from last study treatment) during the study, PFS will be censored at the day of the last tumor assessment. Participants without any post-baseline assessments or with all post-baseline assessments having unknown result/response but known to be alive at the clinical cut off for the analysis will be censored at the date of study treatment initiation plus one day.
Change on CEACAM5 tumor expression levels | Baseline, Cycle 2 Day 2, Discontinuation visit (up to 28 months)
  Mandatory for the 4th-12th participant of each dose level
Change on CEA tumor expression levels | Baseline, Cycle 2 Day 2, Discontinuation visit (up to 28 months)
  Mandatory for the 4th-12th participant of each dose level
Change on FAP tumor expression levels | Baseline, Cycle 2 Day 2, Discontinuation visit (up to 28 months)
  Mandatory for the 4th-12th participant of each dose level
Change on 4-1BB tumor expression levels | Baseline, Cycle 2 Day 2, Discontinuation visit (up to 28 months)
  Mandatory for the 4th-12th participant of each dose level

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Rigshospitalet, København Ø, Denmark
- NKI/AvL, Amsterdam, Netherlands
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (7):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Clinica Universidad de Navarra Madrid, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
- United Kingdom (2):
  - Christie Hospital NHS Trust, Manchester
  - Churchill Hospital, Oxford